CLINICAL TRIAL: NCT06964893
Title: The Effect of Early Postoperative Pain on Postoperative Delirium (POD) in Elderly Patients Undergoing Abdominal Surgery:a Secondary Analysis of Multicenter Prospective Data
Brief Title: The Effect of Early Postoperative Pain on Postoperative Delirium (POD) in Elderly Patients Undergoing Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Taihe Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director, Department of Anesthesiology (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-POD-003
Record Dates: First submitted 2025-04-29; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium (POD)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the mild pain group (NRS <4): An NRS score <4 on postoperative day 1 was classified as mild pain
- the moderate-to-severe pain group: An NRS score ≥4 on postoperative day 1 indicated moderate-to-severe pain

SUMMARY:
This research project is an observational cohort study, representing a secondary analysis of multicenter prospective data from China spanning 2020 to 2022. The study aims to investigate the impact of moderate to severe acute pain on the first postoperative day (POD1) on delirium and anxiety and depression states in elderly patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Post operative delirium will be diagnosed using the 3D- CAM(Confusion Assessment Method) which tests for four features with a series of questions. The features include 1) acute onset and fluctuating course,2) inattention,3) disorganized thinking and 4) altered level of consciousness. Diagnosis of delirium is made if features 1 and 2 and either 3 or 4 are present. the investigators collected baseline characteristics and demographic data of the patients, including clinical information in the following areas:(1) Baseline characteristics: age, gender, body mass index (BMI), American Society of Anesthesiologists (ASA) physical status score, smoke, alcohol , preoperative history of chronic pain, and comorbidities (hypertension, diabetes mellitus, coronary artery disease, cerebrovascular disease, hepatic insufficiency, and renal insufficiency).(2) Preoperative laboratory tests (the most recent prior to surgery): hemoglobin (Hb), white blood cell count, and serum albumin.(3) Preoperative psychological assessments: anxiety and depression state evaluations.(4) Intraoperative variables: grade of operation, type of surgery, duration of surgery, blood transfusion, blood loss, intraoperative dexmedetomidine and nonsteroidal anti-inflammatory drugs (NSAIDs), drain, and PCIA.In this study, the investigators defined the presence or absence of moderate-to-severe pain on POD1 as the exposure variable, assessed using the Numerical Rating Scale (NRS). An NRS score <4 on POD1 was classified as mild pain, while a score ≥4 indicated moderate-to-severe pain 8. Based on this exposure variable, patients were stratified into two groups: the mild pain group (NRS <4) and the moderate-to-severe pain group (NRS ≥4).The investigators summarized patient characteristics based on the presence or absence of moderate-to-severe pain. Continuous variables were expressed as mean ± standard deviation or median (interquartile range) and compared using t-tests or Mann-Whitney U tests. Categorical variables were presented as frequencies and percentages and compared using chi-square tests. Univariate and multivariate regression models were employed to examine the relationship between early postoperative acute pain and the incidence of POD . Furthermore, propensity score matching and subgroup analyses were conducted to further explore the association between the two.

ELIGIBILITY:
Inclusion Criteria:

1. ≥65 years;
2. Absence of hearing, visual, or cognitive impairments (operationally defined as a Chinese version of the Mini-Mental State Examination [MMSE] score ≤17);
3. Scheduled for elective abdominal surgery;
4. Under general anesthesia with endotracheal intubation;
5. Completion of postoperative delirium, anxiety, and depression assessments.

Exclusion Criteria:

1. History of severe psychiatric disorders or chronic use of psychotropic medications;
2. Surgery performed via natural orifice transluminal endoscopic surgery (NOTES) approach;
3. Undergoing vascular interventional procedures;postoperative transfer to the intensive care unit (ICU);
4. Death within 7 days after surgery. -

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients (≥65 years) scheduled for elective abdominal surgery under general anesthesia with endotracheal intubation, without hearing, visual, or cognitive impairments, who completed assessments for postoperative delirium, anxiety, and depression.
Sampling Method: Probability Sample
Enrollment: 3389 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | within 7 days after surgery
  The incidence of postoperative delirium was assessed by a 3-minute diagnostic interview in the surgical ward (3D-CAM).
Subtype of delirium episodes | within 7 days after surgery
  Confusion Assessment Method (CAM) to assess the subtype of postoperative delirium, including four features: acute change or fluctuation course of mental status; inattention; altered level of consciousness; disorganized thinking.

SECONDARY OUTCOMES:
Incidence of anxiety state | within 7 days postoperatively
  Trained assessors evaluated postoperative anxiety using the Generalized Anxiety Disorder-7 (GAD-7) scale 10,administered at the patient's bedside during the recovery period. A score > 5 was defined as indicating anxiety symptoms.
  These psychological assessments were conducted once during the postoperative hospitalization period, scheduled between postoperative days 3-7. For patients discharged before completing all assessments ( anxiety, or depression), trained researchers performed standardized telephone follow-up evaluations using the same assessment protocols.
Incidence of depression state | within 7 days postoperatively
  Postoperative depressive symptoms were assessed by trained researchers using the validated Chinese version of the Patient Health Questionnaire-9 (PHQ-9) . A score > 5 was defined as indicating depressive symptoms. These psychological assessments were conducted once during the postoperative hospitalization period, scheduled between postoperative days 3-7. For patients discharged before completing all assessments ( anxiety, or depression), trained researchers performed standardized telephone follow-up evaluations using the same assessment protocols.
Classification of postoperative anxiety state | within 7 days postoperatively
  Trained assessors evaluated postoperative anxiety using the Generalized Anxiety Disorder-7 (GAD-7) scale 10,administered at the patient's bedside during the recovery period. A score of 5-8 indicating mild symptoms, 9-14 representing moderate anxiety, and 15-21 reflecting severe anxiety.
Classification of postoperative depression state | within 7 days postoperatively
  Postoperative depressive symptoms were assessed by trained researchers using the validated Chinese version of the Patient Health Questionnaire-9 (PHQ-9) . A score of 5-9 representing mild symptoms and 10-14 indicating moderate symptoms, 15-27 was classified as moderate-to-severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma HY, Lv XC, Zhang C, Zhang ZN, Hao XY, Liu YH, Cao JB, Mi WD, Tong L, Fu Q. The effect of early postoperative acute pain on postoperative delirium in older persons undergoing abdominal surgery: a secondary analysis of multicenter prospective data. Eur Geriatr Med. 2025 Dec 2. doi: 10.1007/s41999-025-01367-w. Online ahead of print. PMID 41329455